CLINICAL TRIAL: NCT02404649
Title: A Prospective Clinical Trial Comparing Conventional Dental Implants and Trabecular Metal™ Dental Implants After Staged Sinus Floor Elevation Procedures
Brief Title: Comparing Conventional Dental Implants and Trabecular Metal™ Dental Implants After Sinus Floor Elevation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Kevin Guze, Clinical Instructor, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HarvardMS
Record Dates: First submitted 2015-03-17; First posted 2015-03-31 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Atrophy of Edentulous Alveolar Ridge; Partial Edentulism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bone Augmention (Active Comparator): Two implant designs in a Sinus Bone Augmentation Procedure. Sinus bone augmentation with Puros Cortico-Cancellous Particulate Allograft (70% Cortico and 30% Cancelleous) (Zimmer Dental- Carlsbad, CA, USA)- one implant will be TMDI (Zimmer Dental- Carlsbad, CA, USA) and the second will be Tapered Screw-Vent TSV-MTX (Zimmer Dental- Carlsbad, CA,USA). Implant stability will be determined by the initial insertion torque and RFV values at time of implant placement and after 1 month of healing on a monthly basis up until 12 months post implant placement.
  Interventions: Device: Two implant designs in a Sinus Bone Augmentation Procedure
- Sinus elevation only (Active Comparator): Two implant designs in a Sinus Floor Elevation Procedure. Placement of two dental implants as mentioned above in sinus bone augmentation by sinus elevation procedure, blood clot and CopiOs Pericardium Membrane (Zimmer Dental- Carlsbad, CA, USA) only. One implant will be TMDI (Zimmer Dental- Carlsbad, CA, USA) and the second will be Tapered Screw-Vent TSV-MTX (Zimmer Dental- Carlsbad, CA,USA). Implant stability will be determined by the insertion torque and RFV values at time of implant placement and after 1 month of healing on a monthly basis up until 12 months post implant placement.
  Interventions: Device: Two implant designs in a Sinus Floor Elevation Procedure

INTERVENTIONS:
Device: Two implant designs in a Sinus Bone Augmentation Procedure — Comparing TMDI (Zimmer Dental- Carlsbad, CA, USA) and Tapered Screw-Vent TSV-MTX (Zimmer Dental- Carlsbad, CA,USA) biological behavior after a sinus bone augmentation procedure.
  Arms: Bone Augmention
Device: Two implant designs in a Sinus Floor Elevation Procedure — Comparing TMDI (Zimmer Dental- Carlsbad, CA, USA) and Tapered Screw-Vent TSV-MTX (Zimmer Dental- Carlsbad, CA,USA) biological behavior after a sinus elevation only procedure.
  Arms: Sinus elevation only

SUMMARY:
This is a research study to test the clinical outcome of Trabecular Metal™ Dental Implants (TMDI) (Zimmer Dental Inc Carlsbad, CA, US) in the Maxillary Sinus region. This project will enroll 30 active subjects who will receive two dental implants in the edentulous maxillary molar region. This 24-month research study will examine the clinical stability of TMDI in both sinus elevation and sinus augmentation environments. The proposed research lays the foundation for improved health care by providing surgeons and restorative dentists with data for determining the effects TMDI have on clinical success in less than optimal osseous environments. The rationale that underlies the investigation is that identification of the influences of trabecular surface design on implant stability in varying bone types will allow routine, predictable use of early loading, which, in turn, will translate into more rapid, economical health care, and improved psychosocial well-being of the patient. If these hypotheses are correct, the results are expected to provide evidence based research data to support early loading and immediate loading of single implants in sites of adequate bone volume, and density with or without the use of graft materials in sinus lift procedures. In addition, it is expected that these results will fundamentally advance the field of implant dentistry and bioengineering by providing information on the principles of the bone density-mechanical environment-implant stability interaction.

DETAILED DESCRIPTION:
Specific Aims

Primary Outcome Measures:

• The objective of this study is to allow a preliminary analysis of the resonance frequency values over the 12 month period, which will be the primary outcome

Secondary Outcome Measures:

• To assess Crestal bone level maintenance

Study Arms Bone Augmentation: Placement of two dental implants in Sinus augmented with Puros Cortico-Cancellous Particulate Allograft (70% Cortico and 30% Cancelleous) (Zimmer Dental- Carlsbad, CA, USA)- one implant will be TMDI (Zimmer Dental- Carlsbad, CA, USA) and the second will be Tapered Screw-Vent TSV-MTX (Zimmer Dental- Carlsbad, CA,USA). Implant stability will be determined by the initial insertion torque and RFV values at time of implant placement and after 1 month of healing on a monthly basis up until 12 months post implant placement.

Sinus Elevation only: Placement of two dental implants as mentioned above in sinus augmented by sinus elevation procedure, blood clot and CopiOs Pericardium Membrane (Zimmer Dental- Carlsbad, CA, USA) only. One implant will be TMDI (Zimmer Dental- Carlsbad, CA, USA) and the second will be Tapered Screw-Vent TSV-MTX (Zimmer Dental- Carlsbad, CA,USA). Implant stability will be determined by the insertion torque and RFV values at time of implant placement and after 1 month of healing on a monthly basis up until 12 months post implant placement.

ELIGIBILITY:
Inclusion Criteria:

* • The subject male or female between 21-75 years of age and has:

  * The ability to understand and sign the informed consent prior to starting the study
  * The ability and willingness to comply with all study requirements
  * Adequate oral hygiene
  * The presence of a atrophic, pneumatized, partially edentulous maxilla requiring a lateral approach technique
  * Adequate bone volume to accommodate the planned endosseous dental implant (e.g. sufficient height of bone (5 mm or greater) such that the implant would achieve primary stability, and sufficient width that the implant could be placed within the confines of the existing bone without dehiscence or fenestration. The only implant length utilized in this protocol will be a 10 mm long TMDI (Zimmer)
  * Existing teeth that are healthy and adequately restored, and desired a fixed restoration on implants
  * had a negative pregnancy test within one week prior to surgery, if of childbearing potential.

Exclusion Criteria:

* Subjects who have smoked cigarettes or chewed tobacco within the past year
* History of alcoholism or drug abuse within the past 5 years
* Subjects with Severe bruxing or clenching habits
* Untreated periodontitis
* Subjects at undue risk for an outpatient surgical procedure
* Subjects with the presence of residual roots at the implant site
* Subjects with history of site development (extensive bone augmentation) at the implant site in the past 4 months
* Placement of implant in an extraction site that had been healing for less than 2 month
* Presence of local inflammation or mucosal diseases such as lichen planus
* Subjects with uncontrolled diabetes (defined as HA1c > 7.0 percent)
* Subjects with current hematologic disorder or chronic use of Coumadin (or similar) anti-coagulant therapies
* Subjects with history of leukocyte dysfunction and deficiencies
* Subjects with Metabolic bone disorders
* Subjects with history of renal failure
* Subjects with history of liver disease
* Immunocompromised Subjects having HIV, RA, SLE or other collagen vascular disorders
* Subjects with chronic corticosteroid use
* Subjects undergoing chemotherapy
* Subjects with a history of use of IV-based bisphosphonates
* Subjects with history of radiation treatment to the head or neck
* Subjects requiring grafting of bone or mucosal tissue at the time of implant placement, which would require submersion of the implant during the healing period
* Subjects using of any investigational drug or device within the 30 day period immediately prior to implant surgery
* Pregnant women or women intending to become pregnant during this study period.
* Subjects requiring submersion of implants for esthetic reasons

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-07; Primary Completion 2014-10 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Guze, DMD DMSc MSc, Principal Investigator — Harvard School of Medicine
Locations (1):
- Harvard School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of patients were fulfilled in a timely manner. Patients were were down from the existing patient pool at the Harvard School of Dental medicine.
Pre-assignment Details: Three participants were excluded from the trial due to early dental implant failures. These three events were caused by local infections and thus subsequent readings were not taken.
Groups:
- Bone Augmention: Placement of two dental implants in Sinus augmented with Puros Cortico-Cancellous Particulate Allograft (70% Cortico and 30% Cancelleous) (Zimmer Dental- Carlsbad, CA, USA)- one implant will be TMDI (Zimmer Dental- Carlsbad, CA, USA) and the second will be Tapered Screw-Vent TSV-MTX (Zimmer Dental- Carlsbad, CA,USA). Implant stability will be determined by the initial insertion torque and RFV values at time of implant placement and after 1 month of healing on a monthly basis up until 12 months post implant placement. Thickness of bone surrounding implant body positioned in the sinus will be measured.
  Comparing Conventional Dental Implants and Trabecular Metal™ Dental Implants (Zimmer) after Staged Sinus Bone Augmentation Procedures: Comparing conventional implant versus trabecular metal implant biological behavior in a sinus bone augmentation environment.
  sinus bone augmentation
- Sinus Elevation Only: Placement of two dental implants as mentioned above in sinus augmented by sinus elevation procedure, blood clot and CopiOs Pericardium Membrane (Zimmer Dental- Carlsbad, CA, USA) only. One implant will be TMDI (Zimmer Dental- Carlsbad, CA, USA) and the second will be Tapered Screw-Vent TSV-MTX (Zimmer Dental- Carlsbad, CA,USA). Implant stability will be determined by the insertion torque and RFV values at time of implant placement and after 1 month of healing on a monthly basis up until 12 months post implant placement. Thickness of bone surrounding implant body positioned in the sinus will be measured.
  Comparing Conventional Dental Implants and Trabecular Metal™ Dental Implants (Zimmer) after Staged Sinus Floor Elevation Procedures: Comparing conventional implant versus trabecular metal implant biological behavior in a sinus elevation only environment.
  sinus elevation only
Period: Overall Study
Arm/Group | Bone Augmention | Sinus Elevation Only
Started | 17 | 16
Completed | 16 | 14
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Population: Units: participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Bone Augmention | Sinus Elevation Only | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Resonance Frequency Values of Dental Implants
Description: Implant stability quotient (ISQ) is the value on a scale that indicates the level of stability and osseointegration in dental implants. The scale ranges from 1 to 100 and is measured by implant stability meters instruments using resonance frequency analysis (RFA) technique. The acceptable stability range lies between 55-85 ISQ. Lower initial stability will normally increase with time due to the lower mechanical stability being enforced by the bone remodeling process (osseointegration). The overall average ISQ value of all implants over time is approximately 70. A significant decrease in ISQ indicates a potential problem and should be considered an early warning. For each time period three measurements were taken from three different positions on the dental implant and the measurements were averaged for each time period.
Time Frame: 8 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bone Augmention | Sinus Elevation Only
Number analyzed (Participants) | 16 | 14
units on a scale | 83.04 (3.94) | 80.59 (7.69)

2. Secondary Outcome: Crestal Bone Levels
Description: Evaluating crestal bone levels were performed by measuring (millimeters) vertical bone height gain in the maxillary 2 years postoperatively from CBCT images between control and test group.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Bone Augmention | Sinus Elevation Only
Number analyzed (Participants) | 13 | 11
millimeters | 13.05 (1.73) | 11.68 (1.4)

ADVERSE EVENTS:
Arm/Group | Bone Augmention | Sinus Elevation Only
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less